CLINICAL TRIAL: NCT05142059
Title: Fall Risk Assessment in a Population of Charcot-Marie-Tooth Disease Type 1A (CMT 1A) by Timed Up and Go Test
Acronym: DeteCTCMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2020 REYNAUD 2; 2020-A00344-35 (Other: ANSM)
Record Dates: First submitted 2021-10-12; First posted 2021-12-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Charcot-Marie-Tooth Type 1A Neuropathy
Keywords: Charcot-Marie-Tooth disease type 1A neuropathy; Fall risk; Walking; Timed Up and Go test; 6-Minutes Walk test
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Intervention Model Description: The patients will be recruited in the PMR and neurology departments within the framework of their pathology (current care) and via an older cohort of CMT1A. During a follow-up medical consultation, patients will be informed about the study. If patients express an interest, participants will be listed as a potential attendee. After reflection, patients will be contacted to confirm their participation and an appointment will be set. An assessment will be carried out within the PMR Department of Clermont-Ferrand University Hospital. The doctor will present the protocol in detail to the patients. Upon reading the information form, the doctor will obtain written consent. Clinical information and the results of the various tests will be recorded. Participants will then be compared with each other and over time. Secondly, patients will be contacted by telephone at 6 months to receive any self-reported fall via a standardized questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental cohort (Experimental): Participants will be involved in an evaluation program combining physical tests and self-administered questionnaires. Participants will be followed for 1 year with evaluations taking place at 6 months (occurrence of a fall) and at 1 year (the same evaluation, as initial).
  Interventions: Diagnostic Test: Exploratory physiopathology study, including non-invasive functional explorations carried out in patients with Charcot-Marie-Tooth disease type 1A

INTERVENTIONS:
Diagnostic Test: Exploratory physiopathology study, including non-invasive functional explorations carried out in patients with Charcot-Marie-Tooth disease type 1A — The data of the gait analysis, posturography and strength analyses as well as the questionnaires' scores will be taken into account in this research. At 6 months and at 1 year, occurrence of a fall will be recorded in order to prospectively monitor this parameter. A final analysis will be carried out at 1 year from the first according to the same methods as the initial assessment.

SUMMARY:
The main objective of this study is to explore the relationship between the onset of fall and the time taken to complete the Timed Up and Go test (TUG) in this CMT1A patient population.

The investigators hypothesize that patients with balance disorders and therefore a risk of major fall will require a longer time to perform the Timed Up and Go test. In addition, it seems important to confirm that the severity of the disease has a negative impact on the frequency of balance disorders.

DETAILED DESCRIPTION:
Charcot-Marie Tooth disease is the most frequent and common inherited neuropathy with the various forms and subtypes. The CMT-1A is the most frequent form of the disease and represents more than eighty percent of the all subtypes. In view of different clinical elements (muscular strength deficit, walking and balance disorders, podological impairment), patients with CMT seem to be able to present an increased risk of fall. In 2017 pilot study supports this. More recently, a study by Ramdharry et al. appears to confirm this with a cohort of 252 patients with CMT, 86% of whom have experienced at least one major fall or loss of balance. This increased incidence of falls is also found in children and adolescents with CMT with consequences in terms of injury and management.

Systematic screening of the risk of falls in this population is necessary, but no prospective studies on the occurrence of falls and its detection have yet been carried out in this population.

A study focusing on this issue in order to standardize the assessment of postural control disorders using a simple test of common clinical practice seems necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Diagnosis of Charcot Marie Tooth disease, type 1A confirmed by molecular biology (duplication 17.p11.2) and by a pathological electromyogram, that is to say with demyelinating impairment (+/- axonal) dependent length
* Listening and written French
* Strength of the quadriceps superior to 2/5 MMT MRC
* Agreement after written information, clear and honest about the purpose of the study, the nature of the tests and their possible side effects or bothersome
* Health insurance cover

Exclusion Criteria:

* Presence of other neurological comorbidity
* Presence of coronary artery disease unstabilized
* Peripheral neuropathy of other causes: diabetes, monoclonal gammopathy, malignancy, solid cancer, systemic autoimmune disease (lupus, Sjögren's disease, Wegener sarcoidosis ...), infectious disease (viral hepatitis, HIV ...), drugs known to be responsible for iatrogenic neuropathy.
* Gait trouble of other origin
* Patients unable to give their consent.
* Intellectual deficit that does not allow to comply with tests
* Patient under guardianship, or protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Main explanatory variable: Time to complete the Timed Up and Go test (TUG) (in seconds) | 1 day , 6 months, 12 months
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Investigators measures an evolution or not at 6 months and 1 years.
Main dependent variable: Self-reported occurrence of fall. | 6 months , 12 months
  A fall book will be issued to the patient during the first consultation to trace the date, the circumstances of occurrence. Investigators seek to find an improvement or not in the number of falls at 6 months and 1 year.

SECONDARY OUTCOMES:
: Muscle Strength measured by Medical Research Council (MRC) Scale | Day 0 , 12 months
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle. The patient's effort is graded on a scale of 0-5: Grade 5: Muscle contracts normally against full resistance and Grade 0: No movement is observed.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Day 0 , 12 months
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the device.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Day 0 , 12 months
  Maximum voluntary isometric strength of the quadriceps muscles will be measured with the CYBEX device.
Body Mass Index (Kg/m²). | Day 0 , 12 months
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Height (cm). | Day 0 , 12 months
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations.
Weight (Kg). | Day 0 , 12 months
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Sarcopenia risk. | : Day 0 , 12 months
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Coudeyre, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Result] Reilly MM, Shy ME, Muntoni F, Pareyson D. 168th ENMC International Workshop: outcome measures and clinical trials in Charcot-Marie-Tooth disease (CMT). Neuromuscul Disord. 2010 Dec;20(12):839-46. doi: 10.1016/j.nmd.2010.08.001. Epub 2010 Sep 17. No abstract available. PMID 20850975
- [Result] Ramdharry GM, Thornhill A, Mein G, Reilly MM, Marsden JF. Exploring the experience of fatigue in people with Charcot-Marie-Tooth disease. Neuromuscul Disord. 2012 Dec;22 Suppl 3:S208-13. doi: 10.1016/j.nmd.2012.10.016. PMID 23182641
- [Result] Ribiere C, Bernardin M, Sacconi S, Delmont E, Fournier-Mehouas M, Rauscent H, Benchortane M, Staccini P, Lanteri-Minet M, Desnuelle C. Pain assessment in Charcot-Marie-Tooth (CMT) disease. Ann Phys Rehabil Med. 2012 Apr;55(3):160-73. doi: 10.1016/j.rehab.2012.02.005. Epub 2012 Mar 6. English, French. PMID 22475878
- [Result] Reynaud V, Muti D, Pereira B, Greil A, Caillaud D, Richard R, Coudeyre E, Costes F. A TUG Value Longer Than 11 s Predicts Fall Risk at 6-Month in Individuals with COPD. J Clin Med. 2019 Oct 22;8(10):1752. doi: 10.3390/jcm8101752. PMID 31652506
- [Result] Anens E, Emtner M, Hellstrom K. Exploratory study of physical activity in persons with Charcot-Marie-Tooth disease. Arch Phys Med Rehabil. 2015 Feb;96(2):260-8. doi: 10.1016/j.apmr.2014.09.013. Epub 2014 Oct 5. PMID 25286435